CLINICAL TRIAL: NCT03615703
Title: Functional Neuroimaging Study to Validate the Point Subtraction Aggression Paradigm (PSAP) Task in Typically Developing Children (TDC) Aged 8-12 Years
Brief Title: Functional MRI Study in Healthy Children Engaged in Aggressive Behaviors
Status: Completed | Type: Observational
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 810P204a
Record Dates: First submitted 2018-07-24; First posted 2018-08-06 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-02

CONDITIONS: Impulsive Aggression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this non-interventional study is to optimize the point subtraction aggression paradigms (PSAP) task in typically developing children (TDC).

DETAILED DESCRIPTION:
The PSAP is a behavioral aggression test used to evaluate behavioral response related to impulsive aggression. The task will be combined with functional MRI to establish a reliable BOLD signal during testing in developing healthy subjects (8-12 years old) and, to determine the feasibility to perform the task.

Additionally, the levels of neurotransmitters Glutamate and GABA will be measured using magnetic resonance spectroscopy (MRS).

ELIGIBILITY:
Inclusion Criteria:

Healthy male or female subjects, aged 8-12 years (inclusive) at the time of screening.

Exclusion Criteria:

1. Current history of developmental, psychiatric, or neurologic disorder, including seizures (except for uncomplicated brief febrile seizures), tumor, severe head injury/traumatic brain injury, stroke, lesion, or disease.
2. Known or suspected intelligence quotient (IQ) <70, diagnosis of mental retardation or cerebral palsy or speech/language disorder and history of implanted brain stimulator, vagal nerve stimulator, ventriculoperitoneal shunt, cardiac pacemaker, orthodontic braces, or implanted medication port.
3. Visual and hearing (≥25 dB) impairment.
4. Pre-existing medical or psychological conditions that preclude being in the MRI scanner (e.g., claustrophobia, morbid obesity, or marked anxiety about the procedure).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Brain Imaging in typically developing healthy children during the PSAP aggression Task | The study consist of one visit (total time-2 hrs.).
  The study has only one visit (approximately 2 hours). During the task each participant competes against a fictitious opponent (a computer in reality) to earn points. The participant will play a computer game in which they can steal points (simulating an aggressive behavior) or have points stolen by the opponent.
  10 healthy subjects will be recruited for the study. To make the participant feel comfortable in the MRI, eligible subjects will spend time first to habituate to the scanner and then practice the task. The complete MRI will last one and half hour (at most).
  Functional imaging data (neural activation) will be collected during the behavioral aggression task, while playing the game. In addition, imaging data will be collected at resting state to understand the connectivity between regions of interest before and after the aggression task.

SECONDARY OUTCOMES:
GABA and Glutamate Levels | The study consist of one visit (total time-2 hrs.).
  During the MRI scan, imaging data will be obtained while participants are able to listen to music. GABA and Glutamate signals measured using magnetic resonance spectroscopy (MRS) from two brain regions (anterior cingulate cortex and amygdala) will be used to quantify the two neurotransmitters.

CONTACTS AND LOCATIONS:
Locations (1):
- Meridien Research, Inc., Orlando, Florida, United States

REFERENCES:
- [Background] Cherek DR, Moeller FG, Schnapp W, Dougherty DM. Studies of violent and nonviolent male parolees: I. Laboratory and psychometric measurements of aggression. Biol Psychiatry. 1997 Mar 1;41(5):514-22. doi: 10.1016/s0006-3223(96)00059-5. PMID 9046983
- [Background] Bubenzer-Busch S, Herpertz-Dahlmann B, Kuzmanovic B, Gaber TJ, Helmbold K, Ullisch MG, Baurmann D, Eickhoff SB, Fink GR, Zepf FD. Neural correlates of reactive aggression in children with attention-deficit/hyperactivity disorder and comorbid disruptive behaviour disorders. Acta Psychiatr Scand. 2016 Apr;133(4):310-23. doi: 10.1111/acps.12475. Epub 2015 Aug 21. PMID 26292852